CLINICAL TRIAL: NCT03827044
Title: POLEM:Avelumab Plus 5-FU Based Chemotherapy as Adjuvant Treatment for Stage 3 MSI-High or POLE Exonuclease Domain Mutant Colon Cancer: A Phase 3 Randomised Study
Brief Title: Avelumab Plus 5-FU Based Chemotherapy as Adjuvant Treatment for Stage 3 MSI-High or POLE Mutant Colon Cancer
Acronym: POLEM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: POLEM encountered significant recruitment challenges. With little prospect of recruiting to target the decision to close was made.
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University of Surrey (Other); University of Oxford (Other); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4673 POLEM
Record Dates: First submitted 2018-07-26; First posted 2019-02-01 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: POLE Exonuclease Mutant Colon Cancer; Microsatellite Instability; Stage III Colon Cancer
Keywords: colon cancer; dMMR; POLE exonuclease domain mutant
MeSH Terms: conditions — Microsatellite Instability; Colonic Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Avelumab (Experimental): 6 months of 2 weekly Avelumab
  Interventions: Drug: Avelumab
- No intervention (No Intervention): After standard adjuvant 5FU based chemotherapy, patients will have no active intervention but will start standard follow up.

INTERVENTIONS:
Drug: Avelumab — Avelumab is a fully human monoclonal antibody (MoAb) of the immunoglobulin G (IgG) 1 subtype which specifically binds to the PD-L1 cell surface ligand and blocks its interaction with the PD-1 cell surface receptor.
  Other Names: Bavencio
  Arms: Avelumab

SUMMARY:
The purpose of this study is to determine if dMMR and/or POLE exonuclease domain mutant stage III colon cancer patients gain clinical benefit (i.e. improvement in disease free and overall survival) from PD-L1 inhibitors after standard fluoropyrimidine-based adjuvant chemotherapy.

Avelumab binds PD-L1 and blocks the interaction between PD-L1 and PD-1. This removes the suppressive effects of PD-L1 on anti-tumour CD8+ T cells, resulting in the restoration of cytotoxic T cell response.

The rationale of giving Avelumab after standard adjuvant chemotherapy to this well-defined, molecularly-selected, group is based on the fact that dMMR and POLE exonuclease domain mutant CRCs have a highly and ultra-mutated genetic profile, respectively, thus leading to a high number of neo-antigens with associated over expression of immune checkpoint related proteins. This profile is expected to be highly responsive to checkpoint inhibition as suggested by data of PD-1 inhibitors in dMMR/MSI-H metastatic CRCs.

If this study meets the primary endpoint, using Avelumab in the adjuvant setting following standard chemotherapy would become the standard of care for patients with dMMR and/or POLE exonuclease domain mutant colon cancers. Furthermore, given the availability of molecular markers for patient selection, funders of healthcare would be more likely to fund this treatment.

This study also provides a unique opportunity to conduct translational research analyses on pre- and post-treatment tumour tissue samples and blood samples from dMMR or POLE mutant CRC patients treated with the checkpoint inhibitor Avelumab.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, randomised, phase III trial comparing standard fluoropyrimidine based adjuvant chemotherapy followed by Avelumab (experimental arm) with standard fluoropyrimidine-based adjuvant chemotherapy alone (control arm) in patients who have undergone radical surgical resection for stage III dMMR or POLE exonuclease domain mutant colon cancer. Patients will be stratified in a 1:1 ratio for dMMR status, POLE mutation and type of adjuvant chemotherapy (i.e., 24 weeks of single agent capecitabine chemotherapy versus 12 weeks of CAPOX chemotherapy).

According to the statistical design, 402 patients (201 per arm) are to be randomised. It is expected that approximately 4000 participants will need to be screened in order to recruit 402 patients to the study, assuming an incidence of dMMR of 10-15% and an incidence of POLE mutations of 7% in under 50s (unpublished data from Tomlinson group). Considering the time required to obtain local approval and to initiate all participating centres, the study is expected to take up to 36 months to complete accrual.

There are no proscriptive criteria for surgical resection of the primary tumour in this trial. It is however expected that resection of the tumour will be undertaken in the elective setting by a colorectal specialist surgeon.

Tumour MMR status will be routinely tested locally as per NICE guidelines (either in the pre-operative biopsy or resection specimen). Subjects whose tumours are dMMR can sign the main study consent and undergo the study screening procedures. If they are found to fulfil all eligibility criteria, then they will be randomised. Subjects who are below 50 and whose tumours are pMMR, will be asked to sign a prescreening consent for the centralised analysis of POLE exonuclease domain mutations. This will be done at Oxford Molecular Diagnostics Centre, John Radcliffe Hospital, Headington, Oxford. Those who have tumours harbouring these mutations can sign the main study consent and undergo the study screening procedures. If they are found to fulfil all eligibility criteria, then they will be randomised.

All eligible patients who are randomised will receive standard fluoropyrimidine-based adjuvant chemotherapy for 12 or 24 weeks depending on the decision of the local investigator. The choice of adjuvant chemotherapy (i.e., 24 weeks of single agent fluoropyrimidine chemotherapy or 12 weeks of doublet, oxaliplatin-based chemotherapy) must be declared by the investigator at study entry before randomisation. Type of adjuvant chemotherapy (i.e., 24 weeks of single agent capecitabine or 12 weeks of capecitabine plus oxaliplatin). will be used as stratification factor alongside MMR status and POLE mutation.

At the end of adjuvant chemotherapy, patients who are randomised to the investigational arm, will receive additional 24 weeks of treatment with Avelumab.

After completion of treatment, all subjects will be followed up for up to 7 years from the start of adjuvant chemotherapy.

Correlative biomarker analyses will be conducted as part of the translational study in tumour tissue samples from the resection specimens, tumour tissue samples from the relapsed tumour (if applicable, feasible and upon patient consent) and serial blood samples collected at study entry, during adjuvant treatment and follow-up.

*** POLEM encountered significant recruitment challenges. Recruitment into the study was halted at 30 patients enrolled from the original target of 402.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years
2. ECOG PS 0/1
3. Histologically proven, stage III (i.e., any T, N1 or N2, M0) adenocarcinoma of the colon (as defined by the presence of the inferior pole of the tumour above the peritoneal reflection - that is, at least 15 cm from the anal margin).
4. Fully surgically resected tumour with clear resection margins (i.e., >1 mm)
5. Locally confirmed defective mismatch repair (dMMR) tumour (as defined by the lack of staining on either the pre-operative biopsy samples or resection specimens of at least one of the following proteins: MLH1 (mutL homolog 1), MSH2 (mutS homologue 2), MSH6 (mutS homolog 6), PMS2 or centrally confirmed POLE exonuclease domain mutated tumour (in subjects <50 years old with pMMR tumours)
6. Absence of metastases as shown by post-operative CT scan
7. Absence of major post-operative complications or other clinical conditions that, in the opinion of the investigator, would contraindicate adjuvant chemotherapy 8. Adequate hematological function defined by absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet count ≥100 × 109/L, and hemoglobin ≥9 g/dL (blood transfusion before recruitment is allowed)

9. Adequate hepatic function defined by a total bilirubin level ≤1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤2.5 × ULN 10. Adequate renal function defined by an estimated creatinine clearance ≥30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) 11. Negative serum or urine pregnancy test at screening for women of childbearing potential 12. Fertile men and women must agree to take highly effective contraceptive precautions during, and for 6 months after the last dose of chemotherapy or for 1 month after the last dose of Avelumab

Exclusion Criteria:

1. Rectal tumours (as defined by the presence of the inferior pole of the tumour below the peritoneal reflection - that is, <15 cm from the anal margin).
2. Inability to start adjuvant chemotherapy within 12 weeks after surgery
3. Administration of neoadjuvant systemic chemotherapy or radiotherapy before surgical resection of colon cancer
4. Prior organ transplantation, including allogeneic stem-cell transplantation
5. Significant acute or chronic infections including, among others:

   * known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
   * positive test for HBV (Hepatitis B) surface antigen or anti-HCV (Hepatitis C) antibody and confirmatory HCV RNA test
6. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

   * Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
   * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤10 mg/day of prednisone or equivalent
   * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
7. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3 NCI-CTCAE v4.0), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
8. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v4.0; however, alopecia and sensory neuropathy Grade ≤2 is acceptable unless oxaliplatin administration is planned as part of the adjuvant treatment
9. Pregnancy or lactation
10. Known alcohol or drug abuse
11. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
12. Known history of colitis, pneumonitis and pulmonary fibrosis (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment.
13. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
14. Vaccination within 4 weeks of the first dose of Avelumab and while on trial is prohibited except for administration of inactivated vaccines
15. Other invasive malignancy within 2 years except for non-invasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured. Cancer subjects with incidental histological findings of prostate cancer (tumour/node/metastasis stage of T1a or T1b or prostate-specific antigen ˂10) who have not received hormonal treatment may be included, pending a discussion with the study physician.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Primary End point: Disease Free survival | 3 years
  Disease-free survival (DFS) at 3 years. DFS is measured from the date of randomisation to the date of first relapse (radiological or clinical) or death from any cause.

SECONDARY OUTCOMES:
Secondary End Point: Overall Survival | 5 and 7 years
  Overall survival (OS) at 5 and 7 years. OS is measured from the date of randomisation to date of death from any cause.
Secondary End Points: Quality of Life | 5 Years
  Health-related quality of life (HRQoL) quantified by collection of quality of life data using the EORTC QLQ C-30 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire)
Secondary End Points: Toxicity of Investigational Medicinal Product according to the NCI-CTCAE (Common Terminology Criteria for Adverse Events) version 4.0. | 5 Years
  Toxicity according to the NCI-CTCAE (Common Terminology Criteria for Adverse Events) version 4.0.It uses a range of grades from 1 to 5. Specific conditions and symptoms have values for each level, guideline is: 1 - Mild 2 - Moderate 3 - Severe 4 - Life-threatening 5 - Death

CONTACTS AND LOCATIONS:
Overall Officials: Tony Dhillon, Bsc,FRCP, PhD, Principal Investigator — University of Surrey
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau D, Kalaitzaki E, Church DN, Pandha H, Tomlinson I, Annels N, Gerlinger M, Sclafani F, Smith G, Begum R, Crux R, Gillbanks A, Wordsworth S, Chau I, Starling N, Cunningham D, Dhillon T. Rationale and design of the POLEM trial: avelumab plus fluoropyrimidine-based chemotherapy as adjuvant treatment for stage III mismatch repair deficient or POLE exonuclease domain mutant colon cancer: a phase III randomised study. ESMO Open. 2020 Feb;5(1):e000638. doi: 10.1136/esmoopen-2019-000638. PMID 32079623